CLINICAL TRIAL: NCT01732120
Title: Evaluation of the Off-Clamp Robot-Assisted Partial Nephrectomy Technique in the Management of Renal Tumors
Brief Title: Off Clamp Randomization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Midwest Stone Institute. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: myIRB ID 201208091
Record Dates: First submitted 2012-11-16; First posted 2012-11-22 (Estimated); Results first posted 2022-06-09 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-07

CONDITIONS: Renal Cancer; Renal Ischemia
Keywords: off-clamp; partial nephrectomy; renal cancer treatment; renal ischemia
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Off-clamp partial nephrectomy (Experimental): Partial nephrectomy will be performed without clamping of the renal blood vessels.
  Interventions: Procedure: Off-clamp partial nephrectomy
- Traditional partial nephrectomy (No Intervention): Partial nephrectomy will be performed with clamping of the renal blood vessels.

INTERVENTIONS:
Procedure: Off-clamp partial nephrectomy
  Arms: Off-clamp partial nephrectomy

SUMMARY:
The purpose of this research study is to compare the effects on kidney function after performing the removal of a kidney tumor with or without clamping the blood vessels during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and older.
* Patients willing and able to sign consent.
* Patients with an organ confined renal mass planning to undergo a robotic assisted partial nephrectomy (RAPN).
* Patient with Karnofsky Performance Status (KPS) equal to or greater than 40.

Exclusion Criteria:

* Patients under 18.
* Patients with Karnofsky Performance Status (KPS) less than 40.
* Patients with non-organ confined renal masses (invading renal vein, inferior vena cava, peri-renal tissue, ipsilateral adrenal gland, or metastasis).
* Patients with bilateral synchronous renal masses.
* Patients who can not discontinue Plavix, Coumadin or other anti-platelet or anti-coagulant medications.
* Patients with renal lesions determined to be too complex to perform a RAPN without clamp by the surgeon. (The renal mass may be deemed too difficult based on pre-operatively radiological findings. The surgeon's decision to exclude a mass from a robotic assisted partial nephrectomy would be based on a higher risk of positive margin or complication if a RAPN was performed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2017-05-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Figenshau, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Off-clamp Partial Nephrectomy: Partial nephrectomy will be performed without clamping of the renal blood vessels.
  Off-clamp partial nephrectomy
Period: Overall Study
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (9.8) | 59.4 (11.2) | 58.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 29
  Male | 22 | 29 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 37 | 37 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in eGFR
Description: Renal function following nephrectomy with and without clamping will be assessed using: percent change in eGFR from baseline to 3 months post nephrectomy.
Time Frame: baseline and 3 months post nephrectomy
Population: Missing 3 postoperative eGFR from the Traditional Partial Nephrectomy group and 6 from the Off-Clamp Partial Nephrectomy group.
Measure: Mean (95% Confidence Interval); unit: percent change in eGFR
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 34 | 37
percent change in eGFR | -10.7 [-16.1 to -5.3] | -9.4 [-14.0 to -4.8]

2. Primary Outcome: Percent Change From Baseline in Split Renal Function
Description: Renal function following nephrectomy with and without clamping will be assessed using: percent change in split renal function from baseline to 3 months post nephrectomy.
Time Frame: baseline to 3 months post nephrectomy
Population: Missing 1 postoperative renal scan from the Traditional Partial Nephrectomy group and 7 from the Off-Clamp Partial Nephrectomy group.
Measure: Mean (95% Confidence Interval); unit: percent change in split renal function
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 33 | 39
percent change in split renal function | -11.2 [-15.9 to -6.5] | -11.8 [-15.9 to -7.7]

3. Secondary Outcome: Percent of Observations With Positive Surgical Margins.
Description: Oncologic outcomes will be assessed at the time of nephrectomy based on percent of observations with positive surgical margins.
Time Frame: at the time of nephrectomy
Population: Only malignant cases were included in the analysis of positive margins.
Measure: Number (95% Confidence Interval); unit: percent of cases with positive margins
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 32 | 34
percent of cases with positive margins | 6.3 [0.8 to 20.8] | 5.9 [0.7 to 19.7]

4. Secondary Outcome: Estimated Blood Loss
Description: Perioperative outcomes will be assessed based on estimated blood loss at the time of nephrectomy.
Time Frame: At the time of nephrectomy
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 40 | 40
Milliliters | 184.1 (193.3) | 178.5 (207.5)

5. Secondary Outcome: Percent of Observations With Metastasis
Description: Oncologic outcomes will be assessed based on percent of observations with metastasis on follow-up imaging at 3 years post nephrectomy.
Time Frame: 3 years
Population: Only malignant cases were included in the analysis of metastasis on follow-up imaging.
Measure: Number (95% Confidence Interval); unit: percent of cases with metastasis on f/u
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 32 | 34
percent of cases with metastasis on f/u | 0.0 [0.0 to 0.0] | 2.9 [0.1 to 15.3]

6. Secondary Outcome: Operative Time Measured in Minutes.
Description: Perioperative outcomes will be assessed based on operative time measured in minutes at the time of nephrectomy.
Time Frame: At the time of nephrectomy
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 40 | 40
Minutes | 178.0 (44.4) | 156.0 (40.6)

7. Secondary Outcome: Warm Ischemia Time Measured in Minutes.
Description: Perioperative outcomes will be assessed based on warm ischemia time measured in minutes at the time of nephrectomy.
Time Frame: At the time of nephrectomy.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 40 | 40
Minutes | 0.0 (0.0) | 19.1 (7.5)

8. Secondary Outcome: Percent of Observations With Intra-operative Complications.
Description: Perioperative outcomes will be assessed based on percent of observations with intra-operative complications at the time of nephrectomy.
Time Frame: At the time of nephrectomy
Measure: Number (95% Confidence Interval); unit: % of cases with intraop complications
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 40 | 40
% of cases with intraop complications | 2.5 [0.1 to 13.2] | 0.0 [0.0 to 0.0]

9. Secondary Outcome: Number of Hospital Days Post Nephrectomy.
Description: Perioperative outcomes will be assessed based number of hospital days post nephrectomy.
Time Frame: Day of nephrectomy to day of hospital discharge.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 40 | 40
Days | 1.8 (0.9) | 1.7 (1.2)

10. Secondary Outcome: Percent of Observations With Postoperative Complications.
Description: Perioperative outcomes will be assessed based on percent of observations with postoperative complications.
Time Frame: Within 3 months post nephrectomy.
Measure: Number (95% Confidence Interval); unit: % of cases with postop complications
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
Number analyzed (Participants) | 40 | 40
% of cases with postop complications | 20.0 [7.6 to 32.4] | 17.5 [5.7 to 29.3]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from time of study intervention to the three-month post nephrectomy visit.
Arm/Group | Off-clamp Partial Nephrectomy | Traditional Partial Nephrectomy
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/40 | 4/40
Other Adverse Events (participants affected / at risk) | 0/40 | 4/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Off-clamp Partial Nephrectomy (N=40) | Traditional Partial Nephrectomy (N=40)
acute pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
postoperative bleeding (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Off-clamp Partial Nephrectomy (N=40) | Traditional Partial Nephrectomy (N=40)
urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
fever (Infections and infestations) | 0 (0) | 1 (1)
wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT01732120/Prot_SAP_000.pdf